CLINICAL TRIAL: NCT01853163
Title: Exploratory Evaluation of the Potential for Long-term Retention of Gadolinium in the Bones of Patients Who Have Received Gadolinium Based Contrast Agents According to Their Medical History
Brief Title: Long-Term Retention of Gadolinium in Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navitas Life Sciences GmbH (Industry)
Collaborators: Bayer (Industry); GE Healthcare (Industry); Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ALS-Gd64/001
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2020-06

CONDITIONS: Focus: Long-term Retention of Gadolinium-based Contrast Agent
Keywords: Gadolinium; Contrast Agent; Long-term retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GBCA (Other): Patients who have received GBCAs in the past
  Interventions: Procedure: Gadolinium analysis in bone and tissue samples

INTERVENTIONS:
Procedure: Gadolinium analysis in bone and tissue samples — Gadolinium analysis in bone and tissue samples from patients undergoing an orthopaedic surgical procedure who had received GBCAs in the past.

SUMMARY:
The main objective was to prospectively explore the potential for long-term retention of Gadolinium (Gd) in bones in patients who have received a single dose of Gadolinium-based contrast agents (GBCA) or multiple doses of the same GBCA, with moderate or severe renal impairment or stable normal renal function (eGFR > 60 ml/min/1.73 m2) at the time of GBCA injection.

DETAILED DESCRIPTION:
In order to collect additional clinical data this study was requested by the European Medicines Agency to further investigate whether Gd in human bone and skin are detectable for a long time after administration of GBCAs in patients with impaired renal function who had previously received any of the six different contrast agents (Gadobutrol, Gadodiamide, Gadopentetic acid, Gadoteric acid, Gadoversetamide, and Gadoxetic acid) within a magnetic resonance contrast imaging procedure and who are scheduled for an orthopaedic surgical procedure.

For this study the patients have not been administered any GBCA.

Participating sites are located in Germany, Italy, Poland, Spain, Turkey, USA, Japan, India and Republic of Korea.

ELIGIBILITY:
Main Inclusion Criteria:

* Patient scheduled for an orthopaedic surgical procedure
* A minimum of 1 month has elapsed between GBCA dose and scheduled orthopaedic surgical procedure
* Patient belongs to one of the following subgroups with respect to the number of GBCA doses received and the status of their renal function:

  1. patient has stable impaired renal function (at least moderate impairment, eGFR ≤ 60 ml/min/1.73 m2) and has received one GBCA injection at the standard dose (0.025 mmol per kg body weight for Gadoxetic acid and 0.1 mmol per kg body weight for all other agents) or
  2. patient has stable impaired renal function (at least moderate impairment, eGFR ≤ 60 ml/min/1.73 m2) and has received more than one injection of the same GBCA or
  3. patient has stable normal renal function (eGFR > 60 ml/min /1.73 m2) and has received one GBCA injection at the standard dose (0.025 mmol per kg body weight for Gadoxetic acid and 0.1 mmol per kg body weight for all other agents) or
  4. patient has stable normal renal function (eGFR > 60 ml/min/1.73 m2) who have received more than one injection of the same GBCA

Main Exclusion Criteria:

* Patient has received different GBCAs.
* Patient has received intra-articular GBCA or per any other non-i.v. route
* Patient has received any investigational product or has participated in any other clinical trial within 30 days prior to enrolling in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lohmann, Professor MD, Principal Investigator — University Hospital Magdeburg, Germany
Locations (16):
- Cedar-Sinai Medical Center, Los Angeles, California, United States
- Germany (3):
  - University Hospital Halle (Saale), Halle
  - University Hospital Magdeburg, Magdeburg
  - University Hospital Würzburg, Würzburg
- Japan (2):
  - Fukuoka Orthopaedic Hospital, Fukuoka
  - Nissan Tamagawa Hospital, Tokyo
- South Korea (2):
  - Asan Medical Center Orthopedic Surgery, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Spain (3):
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Hospital Vall d'Hebron, Barcelona
  - H.G.U. Gregorio Marañón, Madrid
- Turkey (Türkiye) (5):
  - Koc University Hospital, Orthopaedics and Traumatology Department, Istanbul
  - Acibadem Hospital, Department of Orthopaedics and Traumatology, Istanbul
  - Fatih Sultan Mehmet Training and Research Hospital, Department of Orthopedics and Traumatology, Istanbul
  - Istanbul Sisli Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - Dokuz Eylul University Tıp Faculty, Izmir

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study sample size was decreased on the basis of protocol amendment #2 date 26 FEB 2016.
Groups:
- GBCA Exposure Group - Normal Renal Function.: Patients with normal renal function (eGFR > 60 ml/min /1.73 m2) who received at least one months prior to the scheduled orthopaedic surgical procedure one or multiple injections of the same GBCA.
- GBCA Exposure Group - Impaired Renal Function.: Patients with impaired renal function (eGFR ≤ 60 ml/min/1.73 m2) who received at least one months prior to the scheduled orthopaedic surgical procedure one or multiple injections of the same GBCA.
- GBCA Naive - Control Group With Normal Renal Function.: GBCA naive patients with normal renal function (eGFR > 60 ml/min /1.73 m2)
- GBCA Naive - Control Group With Impaired Renal Function.: GBCA naive patients with impaired renal function (eGFR ≤ 60 ml/min/1.73 m2)
Period: Overall Study
Arm/Group | GBCA Exposure Group - Normal Renal Function. | GBCA Exposure Group - Impaired Renal Function. | GBCA Naive - Control Group With Normal Renal Function. | GBCA Naive - Control Group With Impaired Renal Function.
Started | 45 | 29 | 7 | 11
Completed | 45 | 29 | 7 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GBCA Naive - Control Group With Normal Renal Function.: GBCA naive patients with normal renal function (eGFR > 60 ml/min/1.73 m2)
- Total: Total of all reporting groups
Arm/Group | GBCA Exposure Group - Normal Renal Function. | GBCA Exposure Group - Impaired Renal Function. | GBCA Naive - Control Group With Normal Renal Function. | GBCA Naive - Control Group With Impaired Renal Function. | Total
Number analyzed (Participants) | 45 | 29 | 7 | 11 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.5) | 74.6 (7.37) | 70 (10.88) | 78.4 (5.28) | 69.5 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 2 | 6 | 52
  Male | 21 | 9 | 5 | 5 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 164.1 (11.08) | 158.9 (9.83) | 174 (5.86) | 162.6 (7.58) | 163 (10.63)
Weight [Mean (Standard Deviation); unit: kg] | 76 (21.09) | 66.7 (19.01) | 90 (13.08) | 76.6 (14.86) | 74.2 (20.03)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Total Gadolinium in Trabecular Bone
Description: Concentration of total Gd in trabecular bone determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Population: Note: Below values for both control groups (0 (0%)) are "NA = Descriptive statistics not performed since it does not satisfy 2/3 of GBCA concentration values are available and above BLQ", 2 patients of the control group with impaired renal function have values > BLQ, max 1.921 ug/g.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Groups:
- GBCA Exposure Group - Normal Renal Function: Patients with normal renal function (eGFR > 60 ml/min/1.73 m2) who received at least one months prior to the scheduled orthopaedic surgical procedure one or multiple injections of the same GBCA.
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 0.335 (476.7) | 0.783 (413.8) | 0 (0) | 0 (0)

2. Primary Outcome: Concentration of Total Gadolinium in Cortical Bone
Description: Concentration of total Gd in cortical bone determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Population: Note: Below values for both control groups (0 (0%)) are "NA = Descriptive statistics not performed since it does not satisfy 2/3 of GBCA concentration values are available and above BLQ", 2 patients of the control group with impaired renal function have values > BLQ, max 1.095 ug/g)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 0.298 (467.5) | 0.680 (410.3) | 0 (0) | 0 (0)

3. Secondary Outcome: Concentration of Total Gd in Skin Tissue Samples
Description: Concentration of total Gd in skin tissue samples (determined by ICP-MS (inductively coupled plasma mass spectrometry)), collected at the time of the scheduled orthopaedic surgical procedure, from a biopsy from the edge of the surgical wound or the amputated part. Analysation of a single skin tissue sample; in case of a second surgery a further sample was taken.
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Population: Note: Below values for all groups (0 (0%)) are "NA = Descriptive statistics not performed since it does not satisfy 2/3 of GBCA concentration values are available and above BLQ", 1 patient of the control group with impaired renal function has a value > BLQ, max 0.138 ug/g.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function.
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 0 (0) | 0 (0) | 0 (0) | 0 (0)

4. Secondary Outcome: Concentration of Calcium in Skin Tissue Samples
Description: Concentration of calcium in skin tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function. | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 653.268 (65.9) | 651.478 (55.6) | 474.377 (78.8) | 790.700 (105.8)

5. Secondary Outcome: Concentration of Calcium in Cortical Bone Tissue Samples
Description: Concentration of calcium in cortical bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function. | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 96908.336 (31.8) | 92491.896 (34) | 142662.680 (11.8) | 118447.534 (25.5)

6. Secondary Outcome: Concentrations of Phosphorus in Cortical Bone Tissue Samples
Description: Concentrations of phosphorus in cortical bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function. | GBCA Exposure Group - Impaired Renal Function. | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 52361.735 (30) | 50247.073 (32.1) | 73151.974 (12.7) | 62689.679 (21.6)

7. Secondary Outcome: Concentrations of Sodium in Cortical Bone Tissue Samples
Description: Concentrations of sodium in cortical bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function. | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 5642.001 (22.3) | 5768.821 (19.2) | 5437.226 (15.6) | 5511.498 (28.2)

8. Secondary Outcome: Concentrations of Zinc in Bone Tissue Samples (Cortical)
Description: Concentrations of zinc in cortical bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 78.516 (29) | 79.900 (24.7) | 92.622 (12.1) | 89.539 (19.1)

9. Secondary Outcome: Concentration of Potassium in Cortical Bone Tissue Samples
Description: Concentration of potassium in bone (cortical) tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 488.128 (41.5) | 543.211 (61.9) | 541.822 (51.1) | 426.705 (65.4)

10. Secondary Outcome: Concentrations of Iron in Cortical Bone Tissue Samples
Description: Concentrations of iron in bone (cortical) tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function. | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 38.807 (71.9) | 41.116 (118.9) | 57.069 (88.5) | 32.293 (109.8)

11. Secondary Outcome: Concentration of Calcium in Trabecular Bone Tissue Samples
Description: Concentrations of calcium in trabecular bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 124671.921 (22.2) | 116601.987 (24.2) | 145859.369 (20.3) | 143735.414 (11.5)

12. Secondary Outcome: Concentration of Phosphorus in Trabecular Bone Tissue Samples
Description: Concentrations of phosphorus in bone (trabecular) tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function. | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 65887.298 (17.7) | 62333.483 (18.4) | 74988.227 (20.8) | 74435.230 (11.7)

13. Secondary Outcome: Concentrations of Sodium in Trabecular Bone Tissue Samples
Description: Concentrations of sodium in trabecular bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 4743.199 (19.7) | 4514.245 (19.5) | 4681.874 (13.8) | 4580.294 (14.7)

14. Secondary Outcome: Concentrations of Zinc in Trabecular Bone Tissue Samples
Description: Concentrations of zinc in trabecular bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 83.812 (29) | 85.312 (30.2) | 89.849 (15.4) | 93.524 (18.3)

15. Secondary Outcome: Concentrations of Potassium in Trabecular Bone Tissue Samples
Description: Concentrations of potassium in trabecular bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 42 | 25 | 6 | 9
micrograms/gram | 394.953 (57.2) | 461.425 (81.9) | 679.490 (85.8) | 340.698 (48.6)

16. Secondary Outcome: Concentrations of Iron in Trabecular Bone Tissue Samples
Description: Concentrations of iron in trabecular bone tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 40.142 (96.8) | 42.889 (116.9) | 62.371 (180.5) | 23.709 (68.7)

17. Secondary Outcome: Concentrations of Phosphorus in Skin Tissue Samples
Description: Concentrations of phosphorus in skin tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 1023.978 (36.9) | 1038.525 (32.2) | 1075.359 (34.1) | 1129.268 (52.7)

18. Secondary Outcome: Concentrations of Sodium in Skin Tissue Samples
Description: Concentrations of sodium in skin tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 3711.129 (42.5) | 4146.187 (49.9) | 4660.517 (36.6) | 4871.197 (42.9)

19. Secondary Outcome: Concentrations of Zinc in Skin Tissue Samples
Description: Concentrations of zinc in skin tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 24.639 (59.5) | 28.767 (55.7) | 27.692 (112.3) | 23.537 (32.9)

20. Secondary Outcome: Concentration of Potassium in Skin Tissue Samples
Description: Concentration of potassium in skin tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 1011.939 (41.7) | 1132.855 (45.1) | 1418.726 (31.8) | 1121.846 (34.4)

21. Secondary Outcome: Concentration of Iron in Skin Tissue Samples
Description: Concentration of iron in skin tissue samples determined by ICP-MS
Time Frame: Day 0 (visit 2, surgery); optional visit 6 (second surgery)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/gram
Arm/Group | GBCA Exposure Group - Normal Renal Function | GBCA Exposure Group - Impaired Renal Function | GBCA Naive - Control Group With Normal Renal Function | GBCA Naive - Control Group With Impaired Renal Function
Number analyzed (Participants) | 45 | 29 | 7 | 11
micrograms/gram | 69.452 (86.4) | 103.432 (101.8) | 145.362 (36.4) | 99.477 (79.2)

ADVERSE EVENTS:
Time Frame: Any AE occurring while a patient was in the study (from informed consent until follow-up visit 2 (visit 4 in case of second surgery) taking place approximately within 10-14 days post-surgery).
Groups:
- GBCA Exposure Group: Patients who received at least one months prior to the scheduled orthopaedic surgical procedure one or multiple injections of the same GBCA.
- GBCA Naive Control Group: GBCA naive patients
Arm/Group | GBCA Exposure Group | GBCA Naive Control Group
All-Cause Mortality (participants affected / at risk) | 2/74 | 0/18
Serious Adverse Events (participants affected / at risk) | 3/74 | 2/18
Other Adverse Events (participants affected / at risk) | 35/74 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBCA Exposure Group (N=74) | GBCA Naive Control Group (N=18)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nephrogenic Systemic Fibrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) — In one subject skin biopsy was assessed as "suspicious for NSF". However, there was no clinical evidence for NSF.
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBCA Exposure Group (N=74) | GBCA Naive Control Group (N=18)
Cardiac disorder (Cardiac disorders) | 1 (2) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 13 (15) | 2 (2)
General Disorders And Administration (General disorders) | 8 (10) | 1 (1)
Infections And Infestations (Infections and infestations) | 5 (6) | 2 (2)
Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 12 (13) | 4 (4)
Investigations (Investigations) | 5 (20) | 0 (0)
Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 9 (10) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 2 (2) | 1 (1)
Psychiatric Disorders (Psychiatric disorders) | 11 (12) | 3 (3)
Renal And Urinary Disorders (Renal and urinary disorders) | 2 (2) | 2 (2)
Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Vascular Disorders (Vascular disorders) | 10 (14) | 2 (2)
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 (0) | 2 (3)

LIMITATIONS AND CAVEATS:
Due to EMA recommendation in July 2017 to restrict the use of linear gadolinium based contrast agents in body scans, the enrollment of impaired renal patients with a history of linear GdCA was restricted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT01853163/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT01853163/SAP_001.pdf